CLINICAL TRIAL: NCT02050269
Title: Measuring the Plasma Clearance of Iohexol to Estimate Glomerular Filtration Rate in Intensive Care Unit Patients: Preliminary Feasibility Study
Acronym: IoxRea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO13-SE / IoxRea; 2013-003936-65 (EudraCT Number); 2013-R49 (Other: CPP); 131229A-11 (Other: ANSM)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-10

CONDITIONS: Acute Circulatory Failure
MeSH Terms: conditions — Shock | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iohexol (Experimental): injection of 5 ml of iohexol
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Iohexol, 300 mg/mL

SUMMARY:
The objective of this study is to assess the feasibility of estimating the clearance of iohexol as an indirect measure of glomerular filtration rate in patients with unstable renal function in the intensive care unit through analysis of rich iohexol plasma kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient admitted to intensive care for less than 12 hours
* Acute circulatory failure
* Patient carrying an arterial catheter
* Informed consent obtained
* Affiliated to social security system

Exclusion Criteria:

* Administration of iohexol the week before intensive care admission
* Administration of iohexol expected within 24 hours of study entry
* Known history of cutaneous immediate or delayed allergic reaction to the injection of the product
* Indication for albumin transfusion within 24 hours of potential inclusion in the study
* Pregnancy or breastfeeding in progress
* Patient under guardianship or judicial protection known at the time of inclusion
* Withdrawal of consent
* Administration of iohexol outside the study within 24 hours after administration of iohexol in the context of the study
* Administration of intravenous albumin in the 24 hours following administration of iohexol in the context of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma clearance of iohexol | 24 hours

SECONDARY OUTCOMES:
Plasma clearance of iohexol in patients developping or not acute kidney injury | 7 days
Link between plasma iohexol clearance and kindney injury markers | 24 hours
Link between injury and/or functional kidney dammage and subsequent acute kidney injury | 7 days
Link between plasma iohexol clearance and urinary metabolomic markers | 24 hours
Comparaison of plasma iohexol clearance measured with 3 and 6 vs. 9 kinetic points | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephan EHRMANN, MCU-PH, Principal Investigator — University Hospital, Tours
Locations (3):
- France (3):
  - Hospital La SOURCE, Orléans
  - University Hospital Strasbourg, Strasbourg
  - Service de Réanimation Polyvalente, CHRU de Tours, Tours

REFERENCES:
- [Result] Salmon-Gandonniere C, Benz-de Bretagne I, Mercier E, Joret A, Halimi JM, Ehrmann S, Barin-Le Guellec C. Iohexol clearance in unstable critically ill patients: a tool to assess glomerular filtration rate. Clin Chem Lab Med. 2016 Nov 1;54(11):1777-1786. doi: 10.1515/cclm-2015-1202. PMID 27166722
- [Derived] Desgrouas M, Merdji H, Bretagnol A, Barin-Le Guellec C, Halimi JM, Ehrmann S, Salmon Gandonniere C. Kinetic Glomerular Filtration Rate Equations in Patients With Shock: Comparison With the Iohexol-Based Gold-Standard Method. Crit Care Med. 2021 Aug 1;49(8):e761-e770. doi: 10.1097/CCM.0000000000004946. PMID 33710029